CLINICAL TRIAL: NCT05126979
Title: Study of the Reactogenicity, Safety and Immunogenicity of Flu-M Inactivated Split Influenza Vaccine in Volunteers Aged 18-60 Years
Brief Title: The Objectives of This Study Are Study of the Reactogenicity, Safety and Immunogenicity of Flu-M Inactivated Split Influenza Vaccine in Volunteers Aged 18-60 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMV-VGIR-1-001/15
Record Dates: First submitted 2021-09-28; First posted 2021-11-19 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-10

CONDITIONS: Influenza
Keywords: influenza; flu; vaccine; Flu-M
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flu-M (without a preservative) (Experimental): 15 volunteers were treated with the Flu-M inactivated split influenza vaccine without a preservative
  Interventions: Biological: Inactivated Split Influenza Vaccine
- Flu-M (with a preservative) (Experimental): 15 volunteers were treated with the Flu-M inactivated split influenza vaccine with a preservative
  Interventions: Biological: Inactivated Split Influenza Vaccine
- Placebo (Placebo Comparator): 15 volunteers were treated with a placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Inactivated Split Influenza Vaccine
  Arms: Flu-M (with a preservative); Flu-M (without a preservative)
Biological: Placebo
  Arms: Placebo

SUMMARY:
Study of the Reactogenicity, Safety and Immunogenicity of Flu-M Inactivated Split Influenza Vaccine in Volunteers Aged 18-60 Years

DETAILED DESCRIPTION:
All subjects will be followed up for 21 days post-randomization. The subjects will further be assessed at 2 days, 7 days, 21 days following the booster vaccination. Blood samples will be collected for reactogenicity and safety and immunogenicity assessments before injection and 21 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the volunteers to participate in the clinical study;
* Healthy volunteers (men and women) aged 18-60 years;
* Volunteers with a titer of antibodies to A(H1N1), A(H3N2) and B influenza viruses less than 1:40 in a HI test
* Volunteers able to fulfill requirements of the protocol (i.e. fill out the patient's diary, come to follow-up visits);
* Female participants were obliged to have negative pregnancy test results and use contraceptives throughout the follow-up period (complete contraception for women of reproductive age)

Exclusion Criteria:

* Allergic reactions to chicken protein or any previous influenza vaccination;
* Leukemia, cancer or a positive reaction to HIV infection, hepatitis B and C, syphilis in the medical history;
* Volunteers who received immunoglobulin or blood products within the last three months before the study;
* Guillain-Barre syndrome (acute polyneuropathy) in the medical history;
* Long-term use (more than 14 days) of immunosuppressants or other immunomodulatory drugs for six months before the study;
* Any confirmed or suspected immunosuppressive or immunodeficiency condition;
* Respiratory, cardiovascular failure, impaired liver or kidney function found during a physical examination or laboratory tests at Visit 1;
* Severe birth defects or serious chronic diseases, including any clinically significant chronic diseases of lungs, kidneys, cardiovascular, nervous system, psychiatric diseases or metabolic disorders, confirmed by medical history or objective examination;
* Volunteers who are (or were) patients of a tuberculosis dispensary and/or narcological dispensary and/or neuropsychiatric dispensary
* acute infectious and/or non-infectious diseases at the time of inclusion in the study;
* Exacerbation of chronic diseases;
* Alcohol abuse and/or use of drugs in the past history;
* Pregnancy and lactation;
* Participation in another clinical study within the last 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2016-05-13 (Actual)

PRIMARY OUTCOMES:
Severity of reported local reactions and their relationship with the vaccination | days 1-7
Severity of reported system reactions and their relationship with the vaccination - during 7 days after the vaccination (the day of vaccination and 6 subsequent days) | days 1-7
Severity of local reactions reported by participants of the study and their relationship with the vaccination | days 8-20
Severity of system reactions reported by participants of the study and their relationship with the vaccination | days 8-20
The measurement physical data at each visit of the trial site by the volunteer | days 1-20

SECONDARY OUTCOMES:
The immunogenicity assessment of the vaccine was carried out by the seroconversion factor | Measurements will be taken at screening, then up to 21 days post-vaccination
The immunogenicity assessment of the vaccine was carried out by Geometric mean titer | Measurements will be taken at screening, then up to 21 days post-vaccination
The immunogenicity assessment of the vaccine was carried out by seroprotection levels | Measurements will be taken at screening, then up to 21 days post-vaccination
The immunogenicity assessment of the vaccine was carried out by seroconversion | Measurements will be taken at screening, then up to 21 days post-vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Perm State Medical University named after academician E.A. Wagner, Perm, Russia